CLINICAL TRIAL: NCT06228365
Title: Efficacy of Digital Sedation Compared With Neuroleptanalgesia in Percutaneous Outpatient Surgery for Superficial Venous Insufficiency
Brief Title: Minimally Invasive Superficial Venous Insufficiency Surgery and Digital Sedation
Acronym: CIMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Vivactis M2Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A01948-37
Record Dates: First submitted 2023-12-14; First posted 2024-01-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Superficial Venous Insufficiency
MeSH Terms: interventions — Neuroleptanalgesia

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, open-label, single-centre study in two parallel groups of 200 patients.
  Maximum duration of patient participation in the study = 2 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual neuroleptanalgesic treatment (Active Comparator): - Group 1: local anaesthesia by tumescence + neuroleptanalgesia
  Interventions: Drug: Neuroleptanalgesia
- use of a device incorporating virtual reality software (Experimental): - Group 2: local anaesthesia by tumescence with virtual reality software
  Interventions: Device: use of a device incorporating virtual reality software

INTERVENTIONS:
Device: use of a device incorporating virtual reality software — use of a device incorporating virtual reality software
  Arms: use of a device incorporating virtual reality software
Drug: Neuroleptanalgesia — Usual neuroleptanalgesic treatment
  Arms: usual neuroleptanalgesic treatment

SUMMARY:
Virtual reality has been shown to reduce the pain experienced during medical procedures.

The aim of this study is to determine to what extent the use of this technique could make it possible to defer the administration of neuroleptanalgesia during the endovenous thermal treatment of superficial varicose veins in addition to local anaesthesia by tumescence.

DETAILED DESCRIPTION:
The main objective of the study is to test the non-inferiority of the effect of sedation by the virtual reality device on the intensity of maximum intraoperative pain compared with the usual neuroleptanalgesic treatment, tolerating a margin of non-inferiority of 0.5 points.Pain will be assessed on an ENS immediately at the end of the surgical procedure.

Prospective, randomised, open-label, single-centre study in two parallel groups of 200 patients.

Maximum duration of patient participation in the study = 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over, who has read and signed the consent form for participation in the study after a reflection period (approximately 1 hour).
* Outpatients with superficial venous insufficiency for which a surgical indication has been given
* Patient requiring sedation associated with local anesthesia

Exclusion Criteria:

* Contraindication to local anesthesia or any of the sedatives used in the protocol
* Hearing or visual impairment contraindicating use of the virtual reality headset
* Pregnant or breast-feeding patients
* Unbalanced epilepsy
* Patients under court protection, guardianship or curatorship
* Patients not affiliated to the French social security system
* Patient unable to understand informed information and/or give written informed consent: dementia, psychosis, disturbed consciousness, non-French-speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity assessed by NRS (numerical rating scale) | Day 1
  The intensity of maximum pain during the surgery will be assessed by numerical rating scale (NRS) graduated from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Level of pre-operative anxiety assessed by the patient using the STAI-Y | Day 0
  The anxiety experienced will be assessed by the patient using the STAI-Y scale (Spielberg State Anxiety Inventory).
Level of post-operative anxiety assessed by the patient using the STAI-Y | Day 1
  The anxiety experienced will be assessed by the patient using the STAI-Y scale (Spielberg State Anxiety Inventory).
treatment administered during the procedure | Day 1
  Nature and quantities of additional sedative treatment administered during the procedure
Pain intensity assessed by NRS (numerical rating scale) | Day 1
  Pain intensity assessed by NRS (numerical rating scale)
Overall patient satisfaction post-opérative assessed by NRS (numerical rating scale) | Day 0
  Overall patient satisfaction will be assessed by NRS (numerical rating scale) graduated from 0 (not at all satisfied) to 10 (completely satisfied).
Overall patient satisfaction day 1 assessed by NRS (numerical rating scale) | Day 1
  Overall patient satisfaction will be assessed by NRS (numerical rating scale) graduated from 0 (not at all satisfied) to 10 (completely satisfied).
Surgery duration | Day 0
  Assessment of the surgery duration
Length of stay in the ICU | Day 1
  Length of stay in the ICU
Length of stay in the hospital | Day 1
  Length of stay in the hospital
Resumption of current activities | Day 1
  Resumption of current activities measured by: YES or NO

CONTACTS AND LOCATIONS:
Overall Officials: Lauranne MATRAY, MD, Principal Investigator — Clinique de l'Union
Locations (2):
- France (2):
  - Clinique de l'Union, Saint-Jean
  - Hôpital Privé de Villeneuve d'Ascq - Ramsay Santé 20 Av. de la Reconnaissance, 59650 Villeneuve-d'Ascq, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: No